CLINICAL TRIAL: NCT03445182
Title: Effectiveness of DentalVibe Comfort System in Reducing Injection Pain and Anxiety During Local Anaesthesia in Paediatric Patients
Brief Title: Effectiveness of DentalVibe in Reducing Injection Pain and Anxiety During Local Anaesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PlovdivMU1
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Pain Management; Local Anaesthesia
Keywords: pain control; paediatric dental patients; local anaesthesia; dentalvibe
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Randomized Intervention Model: Split-mouth assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Local anaesthesia with conventional syringe
  Interventions: Procedure: Local anaesthesia with conventional syringe
- DentalVibe group (Active Comparator): Local anaesthesia with conventional syringe + DentalVibe
  Interventions: Device: Local anaesthesia with conventional syringe + Dentalvibe

INTERVENTIONS:
Procedure: Local anaesthesia with conventional syringe — Buccal infiltration in posterior maxillary region with traditional technique. A 27 gauge short needle is inserted in the mucobuccal fold above the tooth to be anesthetized.
  Local anaesthetic infiltration speed 1ml/min. Drug: Local anaesthetic - Ubistesin - 4% Articaine with adrenaline 1: 200 000 1.7 mL
  Arms: Control group
Device: Local anaesthesia with conventional syringe + Dentalvibe — Buccal infiltration in posterior maxillary region. The tip of the DentalVibe device is placed in the mucobuccal fold above the tooth to be anesthetized. The device is activated for 5 s. A 27 gauge short needle is inserted as close as possible to the inner side of the prong while the vibration is still on.
  Local anaesthetic infiltration speed 1ml/min. After injection the needle is withdrawn and vibration continues for another 5 s.
  Drug: Local anaesthetic - Ubistesin - 4% Articaine with adrenaline 1: 200 000 1.7 mL
  Arms: DentalVibe group

SUMMARY:
The aim of this study is to determine the effectiveness of DentalVibe (DV) in reducing injection pain and anxiety associated with local anaesthesia in paediatric patients.

The clinical trial is a randomized split-mouth assignment. Included patients are 8-12 years old requiring local anesthetic infiltration with conventional syringe (CS) for extraction of two primary maxillary molars bilaterally. Eligible patients undergo two single-visit treatments after CFSS-DS measurement before each, where as DV is allocated to either first or second local anaesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on VAS. Secondary outcome measures: self-reported anxiety during injection on FIS; pain-related behavior according to FLACC scale; heart-rate dynamics; patient preference to local anaesthesia method - CS or CS+DV.

DETAILED DESCRIPTION:
Achieving local anaesthesia in children is one of the critical aspects of pain management.

In recent years, several innovative dental appliances have been developed on the concept to reduce the pain of needle injection by applying pressure, vibration, microoscillations or a combination of them.

Тhe aim of this study is to determine the effectiveness of DentalVibe (DV) in reducing injection pain and anxiety associated with local anaesthesia in paediatric patients.

The clinical trial is a randomized split-mouth assignment. Included patients are healthy positive children 8-12 years old requiring local anesthetic infiltration for extraction of two primary maxillary molars bilaterally.

Eligible patients undergo two single-visit treatments after CFSS-DS measurement of dental fear prior to each. Local anaethetic is delivered through buccal infiltration with conventional syringe, where as DentalVibe Comfort System Injection is allocated to either first or second local anaesthesia procedure. Primary outcome measure will be pain felt during injection, reported by patient on visual analogue scale. Secondary outcome measures: self-reported anxiety during injection on Facial Image Scale; pain-related behavior according to FLACC scale; heart-rate dynamics; patient preference to local anaesthesia method - traditional infiltration or DentalVibe-assisted injection.

ELIGIBILITY:
Exclusion criteria:

* Children who are considered medically compromised or medically complex patients. The absence of disease is confirmed by anamnestic interview with a parent or a care-giver of the child and excludes general acute or chronic disease, cognitive impairment, psychogenic nonepileptic events.
* Patients who are undergoing therapy with neurological, sedative, analgesic and/or anti-inflammatory drugs 7 days prior to treatment.
* Patients with allergy to local anesthetics of the amide group.
* Children, who are first time ever dental patients.

Inclusion criteria:

* Patients, identified as positive or definitely positive through Frankl behavioral rating scale.
* Children, requiring local anaesthesia infiltration for extraction of two primary upper jaw molars bilaterally.
* Indications for extraction of primary molars: over-retention - in case of delayed physiological change and tendency of eruption of the permanent tooth; orthodontic reasons - tooth removed to prevent or correct malocclusion; advanced root resorption and imminent physiological tooth replacement; teeth with a severely damaged clinical crown (from trauma or caries and its complications); teeth with failed pulpotomy, acute or chronic diffuse periodontitis, endangering the germ of the permanent tooth.
* Obtained informed consent from parents or gave-givers to participate in the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Pain felt during injection using visual analogue scale | Immediately after local anaesthetic delivery
  Self-reported pain by the patient immediately after local anaesthesia infiltration using a VAS (visual analogue scale), containing a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, including pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst'). The combination allows children to pick a facial expression, that corresponds with their pain and see a number that matches it.

SECONDARY OUTCOMES:
Pain-related behavior evaluated on the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale | During local anaesthesia procedure
  Evaluated by the outcomes assessor. The FLACC scale has five criteria - Faces, Legs, Activity, Cry, Consolability, which are each assigned a score of 0, 1 or 2. Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain.
Self-reported anxiety during injection evaluated on FIS | Immediately after local anaesthetic delivery
  The Facial Image Scale (FIS) comprises a row of five faces from very unhappy (score 5) to very happy (score 1).
Heart rate dynamics of the patient | Start: in the waiting room, at least 5 minutes before local anaesthesia procedure. End: at least 5 minutes after treatment.
  Patient's left index finger is connected to a portable recording pulse oximeter for children.
Assessment of self-reported dental fear on CFSS-DS questionnaire | Prior to each visit
  Assessment will be performed prior to both visits. The Children's Fear Survey Schedule - Dental Subscale (CFSS-DS) questionnaire consists of 15 items related to different aspects of dental treatment, including fear of injections, scored as follows: Not afraid = 1; a little afraid = 2; fairly afraid = 3; quite afraid = 4; and very afraid = 5. Total score: 15 to 75. Children with CFSS-DS ≥32 are defined as dentally anxious.
Patient preference to local anaesthesia method | One week after second procedure
  One week after the second dental visit, the patient is reached by a phone call and asked: "Which method do you prefer to put your tooth to sleep? With the vibrating device or without it?"

CONTACTS AND LOCATIONS:
Overall Officials: Ani Beltcheva, Study Director — Medical University - Plovdiv, Bulgaria
Locations (1):
- Faculty of Dental Medicine, Medical University - Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veneva E, Cholakova R, Raycheva R, Belcheva A. Efficacy of vibrotactile device DentalVibe in reducing injection pain and anxiety during local anaesthesia in paediatric dental patients: a study protocol for a randomised controlled clinical trial. BMJ Open. 2019 Jul 2;9(7):e029460. doi: 10.1136/bmjopen-2019-029460. PMID 31270121